CLINICAL TRIAL: NCT04901676
Title: A Phase 3, Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Leronlimab in Combination With Standard of Care for Moderately Ill Patients With Coronavirus Disease 2019 (COVID-19) Pneumonia
Brief Title: Leronlimab in Moderately Ill Patients With COVID-19 Pneumonia
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Pending DSMB evaluation
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARO_21_018_001
Record Dates: First submitted 2021-05-24; First posted 2021-05-25 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Pneumonia; Leronlimab
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Leronlimab (Experimental): Leronlimab subcutaneously once a week (up to 4 doses) until hospital discharge. The first dose will be of 700 mg, followed by weekly doses of 350 mg.
  Interventions: Drug: Leronlimab
- Placebo (Placebo Comparator): Placebo subcutaneously once a week (up to 4 doses) until hospital discharge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Leronlimab — Leronlimab 700 mg (first dose) followed by weekly 350 mg
  Arms: Leronlimab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Leronlimab (PRO 140) is a humanized IgG4,k monoclonal antibody (mAb) that recognizes the C-C chemokine receptor type 5 (CCR5). Disruption of the C-C chemokine ligand 5 (CCL5)-CCR5 axis via leronlimab-mediated CCR5 blockade might prevent pulmonary trafficking of pro-inflammatory leukocytes and dampen pathogenic immune activation in coronavirus disease 2019 (COVID-19).

The purpose of the study is to assess the safety and efficacy of leronlimab plus standard of care in patients hospitalized with COVID-19 pneumonia who are not requiring mechanical ventilation or extracorporeal oxygenation (ECMO).

DETAILED DESCRIPTION:
Leronlimab (PRO 140) is a humanized IgG4,k monoclonal antibody (mAb) that recognizes the C-C chemokine receptor type 5 (CCR5). CCR5 is expressed predominantly on T cells but also found on macrophages, dendritic cells, and eosinophils to mediate chemotaxis in response to its cognate ligands that include CCL5 (RANTES), CCL3 (MIP-1α), and CCL4 (MIP-1β). These ligands are integral in the recruitment of these immune cells to inflammatory sites. The immunopathogenesis of COVID-19 likely involves the excessive influx of immune cells into the lung. Disruption of the CCL5-CCR5 axis via leronlimab-mediated CCR5 blockade might prevent pulmonary trafficking of pro-inflammatory leukocytes and dampen pathogenic immune activation in COVID-19.

The purpose of the study is to assess the safety and efficacy of leronlimab plus standard of care in patients hospitalized with COVID-19 pneumonia who are not requiring mechanical ventilation or extracorporeal oxygenation (ECMO).

This is a Phase 3, 2-arm, randomized, double blind, placebo controlled, multicenter study to evaluate the safety and efficacy of leronlimab (PRO 140) as an add on therapy to the institutional standard of care (SoC) for the management of moderately ill patients with COVID-19 pneumonia.

Patients will be randomized in a 1:1 ratio to receive up to four doses of leronlimab (PRO 140) or placebo. Leronlimab (700 mg followed by 350 mg weekly) or placebo will be administered subcutaneously over a 4-week treatment period. No treatments will be administered post-discharge.

The participant will be evaluated on each study day while hospitalized up until and including Day 28. The daily visits will capture clinical status - ordinal scale and the occurrence of adverse events. A complete follow-up assessment will be performed at Days 7, 14, 21, 28, 42 and 60 for those who are hospitalized at these specific timepoints. Follow-up visits can be conducted as telephone or video contact visits, if subject is discharged from the hospital prior to the complete follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females aged ≥ 18 years
2. Moderately ill patients with COVID-19 (defined as Ordinal Scale of 5 or 6): Hospitalized, requiring supplemental oxygen or hospitalized, on non-invasive ventilation or high flow oxygen devices
3. Evidence of pneumonia (pulmonary infiltrates) at chest radiography or computed tomography compatible with COVID-19.
4. Hospitalization for less than 72 hours, receiving standard of care treatment for COVID-19.
5. Laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR).
6. Subject (or legally authorized representative) provides written or oral informed consent prior to initiation of any study procedures.
7. Women of childbearing potential and their partner must agree to use at least one highly effective method of contraception (e.g., hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], intrauterine devices, bilateral tubal occlusion, or sexual abstinence) for the duration of the study.

Exclusion Criteria:

1. Subjects on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
2. Subjects who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible.
3. Inability to provide informed consent (from subject or legally authorized representative) or to comply with test requirements.
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk associated with study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Pregnancy or breast feeding.
6. Subject participating in another study with for an investigational treatment.
7. Suspected or known active systemic bacterial, fungal, or viral infections (with the exception of COVID-19), that may increase the risk for the study participant based on investigator judgement.
8. Participants who are immunocompromised, with known immunodeficiencies, or taking potent immunosuppressive agents (e.g., azathioprine, cyclosporine).
9. Patients with estimated discharge or transfer for other hospital in the first 72 hours of study inclusion.
10. Patients with low probability of survival in the first 48 hours of study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of death or respiratory failure until day 28 | 28 days
  Rates of participants who attain categories 6, 7, or 8 on the eight-category ordinal scale within 28 days
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities and/or requiring home oxygen
  3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  5. Hospitalized, requiring supplemental oxygen
  6. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  7. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  8. Death

SECONDARY OUTCOMES:
Time to clinical recovery | 28 days
  Categories 1, 2 and 3 on a 8-point ordinal scale
Death or intubation until day 28 | 28 days
  Categories 7 or 8 on the eight-point ordinal scale
Proportion of patients clinically recovered | Days 14, 28, 42, and 60
  Categories 1, 2 and 3 on a 8-point ordinal scale
All-cause mortality | Days 14, 28, 42, and 60
Proportion of patients discharged alive | Days 14, 28, 42, and 60
  Categories 1 and 2 on a 8-point ordinal scale
Clinical status | Days 14, 28, 42, and 60
  On a 8 point ordinal scale
Length of hospital stay | 28 days
  days

CONTACTS AND LOCATIONS:
Locations (27):
- Brazil (27):
  - Hospital Vitoria, Vitória, Espírito Santo
  - Clinica São Roque, Ipiaú, Estado de Bahia
  - Instituto de Ensino e Pesquisa do Hospital da Bahia, Salvador, Estado de Bahia
  - Santa Casa de Misericórdia da Bahia - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Santa Casa de Passos, Passos, Minas Gerais
  - Hospital São Lucas Copacabana, Rio de Janeiro, Rio de Janeiro
  - Instituto Atena de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica do Coração, Aracaju, Sergipe
  - Fundação PIO XII, Barretos, São Paulo
  - Irmandade do Sr. Bom Jesus dos Passos da Santa Casa de Misericórdia de Bragança Paulista, Bragança Paulista, São Paulo
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Santa Casa de Santos, Santos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Associação Beneficente Síria - Hospital do Coração (HCor), São Paulo, São Paulo
  - BP Mirante, São Paulo, São Paulo
  - Hospital 9 de Julho, São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Hospital Beneficência Portuguesa, São Paulo, São Paulo
  - Hospital M'Boi Mirim, São Paulo, São Paulo
  - Hospital Santa Paula, São Paulo, São Paulo
  - Santa Casa de Votuporanga, Votuporanga, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo

IPD SHARING:
Plan to Share IPD: No